CLINICAL TRIAL: NCT02707536
Title: Influence of Platelet-Rich Fibrin on Post-extraction Alveolar Ridge Healing/Preservation as a Stand-alone or Adjunct to Particulate Graft: A Clinical, Radiographic and Histological Evaluation
Brief Title: Influence of Platelet-Rich Fibrin on Post-extraction Alveolar Ridge Healing/Preservation as a Stand-alone or Adjunct to Particulate Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sridhar V. K. Eswaran, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-14-0190
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Extraction Socket Healing; Alveolar Ridge Preservation
MeSH Terms: interventions — Prolactin-Releasing Hormone; Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No socket grafting (No Intervention): Extraction with normal socket healing
- Socket grafting with platelet rich fibrin (PRF) alone (Active Comparator): Extraction with socket grafting with platelet rich fibrin (PRF) alone.
  Interventions: Procedure: Socket grafting with PRF
- Socket grafting with bone grafting alone (Active Comparator): Extraction with socket grafting using bone graft (xenograft).
  Interventions: Procedure: Socket grafting with bone graft
- Socket grafting with PRF and bone grafting (Active Comparator): Extraction with socket grafting using PRF combined with bone graft (xenograft).
  Interventions: Procedure: Socket grafting with PRF; Procedure: Socket grafting with bone graft

INTERVENTIONS:
Procedure: Socket grafting with PRF — Extraction with socket grafting using PRF.
  Arms: Socket grafting with PRF and bone grafting; Socket grafting with platelet rich fibrin (PRF) alone
Procedure: Socket grafting with bone graft — Extraction with socket grafting using bone graft.
  Arms: Socket grafting with PRF and bone grafting; Socket grafting with bone grafting alone

SUMMARY:
The goal of this project is to evaluate the influence of platelet rich fibrin (PRF) in extraction socket healing with or without particulate bone graft. The hypothesis of this study is that PRF will enhance the extraction socket healing and new bone formation when compared to extraction sockets grafted without PRF.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age
* Hopeless or non-restorable single non-molar tooth per quadrant with adjacent teeth present
* Maximum of two teeth can qualify per patient.
* The buccal plate must be ≥ 1mm in width with a 4-wall configuration.
* Cases requiring minimal sinus grafting (<3mm)
* Bone grafting limited to the apical portion of the osteotomy site

Exclusion Criteria:

* Exclusion Criteria:
* Untreated periodontal disease, endodontic-periodontal disease and/or caries
* The buccal plate must be ≤ 3mm in width with a 4-wall configuration.
* Patients with uncontrolled or severe systemic disease (Diabetes)
* Patients with medical conditions or taking medication associated with compromised bone healing (Diabetes, Autoimmune Dysfunction, Prolonged Cortisone Therapy, Chemotherapy, or Bisphosphonate Therapy)
* Current Smokers
* Subjects with extensive parafunctional habits (ie; bruxism)
* Subjects who demonstrate inadequate oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in alveolar ridge width (buccal-lingual) | baseline, 3 months
  Baseline is at the time of extraction with or without socket grafting.
Change in alveolar ridge height (apical coronal) | baseline, 3 months
  Baseline is at the time of extraction with or without socket grafting.

SECONDARY OUTCOMES:
Percentage of vital bone in bone core as assessed histology | 3 months
  A bone core will be taken at 3 months after socket grafting.
Percentage of residual bone graft in bone core as assessed histology | 3 months
  A bone core will be taken at 3 months after socket grafting.

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Eswaran, BDS, MS, MSD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston School of Dentistry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No